CLINICAL TRIAL: NCT02205476
Title: A Long-term Efficacy Assessment Following Initial Scar Revision Surgery And Phase 2 Open-label Study To Evaluate Safety Of Re-treatment With Pf-06473871
Brief Title: A Phase 2 Extension Study To Enroll Subjects Who Were Enrolled In B5301001 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: B5301001 study did not meet its predefined efficacy endpoints, the long term follow up study B5301012 was terminated in 1/6/2015. No safety concerns identified.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B5301012; 2014-002703-17 (EudraCT Number)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Hypertrophic Scars Resulting From Prior Breast Scar Revision Surgery
Keywords: Phase 2; open-label; safety; hypertrophic scar revision surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): The number of doses each subject receives will be consistent with number received in protocol B5301001 (Group 1 = 4 doses).
  Interventions: Drug: PF-06473871
- Group 2 (Experimental): The number of doses each subject receives will be consistent with number received in protocol B5301001 (Group 2 = 3 doses).
  Interventions: Drug: PF-06473871

INTERVENTIONS:
Drug: PF-06473871 — Subjects who previously were randomized in B5301001 study will go under a second revision surgery followed by 4 administration of PF-06473871.
  Arms: Group 1
Drug: PF-06473871 — Subjects who previously were randomized in B5301001 study will go under a second revision surgery followed by 3 administration of PF-06473871.
  Arms: Group 2

SUMMARY:
Study is a multicenter, two-part, open-label phase II study in adults, evaluating the safety and long-term efficacy of PF-06473871 one year after surgical revision and treatment with PF-06473871.

ELIGIBILITY:
Inclusion Criteria:

* Subjects previously randomized to Pfizer clinical study B5301001.
* Subjects must be able to tolerate up to a 3 hour scar revision surgery under sedation and local anesthesia.

Exclusion Criteria:

* Pregnant female subject; breastfeeding female subjects; male subjects with partners currently pregnant.
* Any previous history of intolerable adverse reactions to PF-06473871, such as serious adverse events attributed to study drug or having been withdrawn due to AE in prerequisite study B5301001.

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Stephan Baker MD PA, Coral Gables, Florida
  - Bayside Ambulatory Center, Miami, Florida
  - Kavali Plastic Surgery and Skin Renewal Center, Atlanta, Georgia
  - Primeter outpatient surgery center, Atlanta, Georgia
  - Body Aesthetic Research Center, St Louis, Missouri

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5301012&StudyName=A%20Phase%202%20Extension%20Study%20To%20Enroll%20Subjects%20Who%20Were%20Enrolled%20In%20B5301001%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received the treatment in previous study B5301001 (NCT01730339), were enrolled in this study.
Pre-assignment Details: Participants who completed part A of the study had the option to obtain scar revision surgery with PF-06473871 in part B of the study. No participant entered into part B due to premature termination of the study.
Groups:
- Group 1: PF--06473871/Placebo (4* 5 mg/cm): Participants with bilateral hypertrophic scars who received 4 intradermal injections of PF-06473871 at a dose of 5 milligram per linear centimeter (mg/cm) (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast in study B5301001 (NCT01730339) were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery.
- Group 2: PF--06473871/Placebo (3* 5 mg/cm): Participants with bilateral hypertrophic scars who received 3 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5 and 8; and 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5 and 8 on another breast in study B5301001 (NCT01730339) were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery.
Period: Overall Study
Arm/Group | Group 1: PF--06473871/Placebo (4* 5 mg/cm) | Group 2: PF--06473871/Placebo (3* 5 mg/cm)
Started | 7 | 3
Completed | 0 | 0
Not Completed | 7 | 3
Not completed — Study termination by Sponsor | 7 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set included all participants who signed an informed consent and for whom data were collected for Part A of this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: PF--06473871/Placebo (4* 5 mg/cm) | Group 2: PF--06473871/Placebo (3* 5 mg/cm) | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (6.80) | 39.0 (15.13) | 40.2 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician Scar Assessment Using Complete Patient and Observer Scar Assessment Scale (POSAS) at Part A Visit
Description: Physician scar assessment was performed using 10-point POSAS scale. Physician rated each of the items (vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion) for a scar on a score of 1 (normal skin) to 10 (worst scar imaginable).
Time Frame: 52 weeks after initial scar revision surgery in study B5301001
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- Group 1: PF--06473871: 4* 5 mg/cm: Participants with bilateral hypertrophic scars who received 4 intradermal injections of PF06473871 at a dose of 5 mg/cm ( 2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8, and 11 in study B5301001 (NCT01730339) and were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery.
- Group 1: Placebo: 4* 5 mg/cm: Participants with bilateral hypertrophic scars who received 4 intradermal injections of PF-06473871 on one breast and 4 intradermal injections of placebo matched to PF-06473871 on another breast at Week 2, 5, 8, and 11 in study B5301001 (NCT01730339) were assessed for efficacy in the part A of the study, 1 year post their initial scar revision surgery.
- Group 2: PF¬06473871: 3* 5 mg/cm: Participants with bilateral hypertrophic scars who received 3 intradermal injections of PF-06473871 on one breast at Week 2, 5 and 8 in study B5301001 (NCT01730339) were assessed for efficacy in the part A of the study, 1 year post their initial scar revision surgery.
- Group 2: Placebo: 3* 5 mg/cm: Participants with bilateral hypertrophic scars who received 3 intradermal injections of PF-06473871 on one breast and 3 intradermal injections of placebo matched to PF-06473871 on another breast at Week 2, 5 and 8 in study B5301001 (NCT01730339) were assessed for efficacy in the part A of the study, 1 year post their initial scar revision surgery.
Arm/Group | Group 1: PF--06473871: 4* 5 mg/cm | Group 1: Placebo: 4* 5 mg/cm | Group 2: PF¬06473871: 3* 5 mg/cm | Group 2: Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 7 | 7 | 3 | 3
units on scale
  Vascularity | 2.71 (1.496) | 2.71 (1.113) | 1.33 (0.577) | 2.00 (1.000)
  Pigmentation | 3.79 (2.307) | 5.00 (2.517) | 2.00 (1.000) | 3.00 (2.000)
  Thickness | 3.86 (2.478) | 4.64 (2.286) | 2.00 (1.000) | 3.00 (2.000)
  Relief | 4.14 (2.795) | 4.36 (2.358) | 2.00 (1.000) | 3.67 (3.055)
  Pliability | 3.50 (2.693) | 3.93 (2.805) | 1.67 (0.577) | 3.67 (3.055)
  Surface Area | 4.86 (2.193) | 4.57 (2.573) | 2.33 (0.577) | 3.33 (2.517)
  Overall opinion | 4.29 (2.628) | 4.64 (2.561) | 2.00 (1.000) | 3.00 (2.000)

2. Secondary Outcome: Patient Global Assessment Using Overall Opinion of Patient and Observer Scar Assessment Scale (POSAS) at Part A Visit
Description: Patient global assessment was performed using the overall opinion question of the POSAS scale. Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin).
Time Frame: 52 weeks after initial scar revision surgery in study B5301001
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- Group 1: PF-06473871: 4* 5 mg/cm: Participants with bilateral hypertrophic scars who received 4 intradermal injections of PF06473871 at a dose of 5 mg/cm ( 2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8, and 11 in study B5301001 (NCT01730339) and were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery.
- Group 2: PF-06473871: 3* 5 mg/cm: Participants with bilateral hypertrophic scars who received 3 intradermal injections of PF-06473871 on one breast at Week 2, 5 and 8 in study B5301001 (NCT01730339) were assessed for efficacy in the part A of the study, 1 year post their initial scar revision surgery.
Arm/Group | Group 1: PF-06473871: 4* 5 mg/cm | Group 1: Placebo: 4* 5 mg/cm | Group 2: PF-06473871: 3* 5 mg/cm | Group 2: Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 7 | 7 | 3 | 3
units on scale | 7.07 (2.281) | 6.57 (3.552) | 3.00 (1.732) | 4.00 (2.646)

3. Secondary Outcome: Patient-Reported Scar Evaluation Questionnaire (PR-SEQ) Symptom and Appearance Domain Score at Part A Visit
Description: PR-SEQ questionnaire consisted of 30 different attributes of scars that included following four dimensions: appearance (5 attributes), symptoms (3 attributes), bothersomeness (8 attributes), and impacts on the quality of life (physical and emotional wellbeing [14 attributes]). Each question had 5 possible responses: not at all (0), slightly (1), moderately (2), very (3), and extremely (4). Subjects completed an abbreviated version which included only the Symptoms and Appearance dimensions to evaluate treatment outcomes. Each of the item scores were transformed into a 0 to 100 scale. Each dimension score was calculated from averaging the transformed scores (0 to 100 scaled) for specified items. Each domain score ranged from 0 to 100, with higher scores indicating higher severity.
Time Frame: 52 weeks after initial scar revision surgery in study B5301001
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Group 1: PF-06473871: 4* 5 mg/cm | Group 1: Placebo: 4* 5 mg/cm | Group 2: PF¬06473871: 3* 5 mg/cm | Group 2: Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 7 | 7 | 3 | 3
units on scale
  Appearance | 46.79 (28.965) | 49.29 (30.745) | 33.33 (12.583) | 48.33 (41.633)
  Symptoms | 23.21 (24.516) | 9.52 (16.962) | 0.00 (0.000) | 0.00 (0.000)

4. Secondary Outcome: Physician and Participant Photoguide Scar Assessment Scale Score at Part A Visit
Description: Physician and participants rated severity of each scar using a photonumeric guide on a scale ranging from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe).
Time Frame: 52 weeks after initial scar revision surgery in study B5301001
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Group 1: PF-06473871: 4* 5 mg/cm | Group 1: Placebo: 4* 5 mg/cm | Group 2: PF¬06473871: 3* 5 mg/cm | Group 2: Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 7 | 7 | 3 | 3
units on scale
  Physician assessment | 2.64 (1.600) | 3.00 (1.414) | 1.33 (0.577) | 2.33 (1.528)
  Participant assessment | 2.79 (1.577) | 3.14 (1.773) | 1.67 (0.577) | 2.67 (2.082)

5. Primary Outcome: Part B: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Vital signs included pulse rate and systolic blood pressure and diastolic blood pressure.
Time Frame: Part B: Baseline up to Week 15
Population: Data for this outcome measure was not analyzed because part B was not initiated due to early termination of the study during Part A.
Groups:
- Group 1: PF--06473871/Placebo: 4* 5 mg/cm: Participants with bilateral hypertrophic scars who received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast in study B5301001 (NCT01730339) were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery and were planned to receive scar revision surgery in part B of the study.
- Group 2: PF--06473871/Placebo: 3* 5 mg/cm: Participants with bilateral hypertrophic scars who received 3 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5 and 8; and 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5 and 8 on another breast in study B5301001 (NCT01730339) were assessed for efficacy in part A of the study, 1 year post their initial scar revision surgery and were planned to receive scar revision surgery in part B of the study.
Arm/Group | Group 1: PF--06473871/Placebo: 4* 5 mg/cm | Group 2: PF--06473871/Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Clinical Laboratory Abnormalities
Description: Clinical laboratory tests included clinical chemistry (sodium, potassium, chloride, bicarbonate, glucose, blood urea nitrogen (BUN), creatinine, albumin, calcium, total, direct and indirect bilirubin, gamma-glutamyltransferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactic dehydrogenase (LDH), alkaline phosphatase, creatine phosphokinase (CPK), uric acid, amylase and lipase) and hematology (hemoglobin, hematocrit, red blood cell count (RBC), white blood cell count (WBC) with differential, and platelet count) tests to be performed.
Time Frame: Part B: Baseline up to Week 15
Population: as for outcome 5
Arm/Group | Group 1: PF--06473871/Placebo: 4* 5 mg/cm | Group 2: PF--06473871/Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Data for this outcome measure was not analyzed because part B was not initiated due to early termination of the study during Part A.
Time Frame: Part B: Baseline up to Week 15
Population: as for outcome 5
Arm/Group | Group 1: PF--06473871/Placebo: 4* 5 mg/cm | Group 2: PF--06473871/Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Volumetric & Colorimetric Scar Assessment (3D Imaging) at Part A Visit
Description: Three-dimension digital photography was planned to be taken of the participants scars for determination of scar volume, height, and color performed in a subset of selected investigational centers equipped with specialized 3D photographic equipment.
Time Frame: 52 weeks after initial scar revision surgery in study B5301001
Population: The volumetric and colorimetric scar assessments were collected under this protocol but were not analyzed.
Arm/Group | Group 1: PF--06473871: 4* 5 mg/cm | Group 1: Placebo: 4* 5 mg/cm | Group 2: PF¬06473871: 3* 5 mg/cm | Group 2: Placebo: 3* 5 mg/cm
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were planned to be assessed in part B of the study. Part B of study was not initiated due to premature termination during part A of the study.
Arm/Group | Group 1: PF--06473871/Placebo (4* 5 mg/cm) | Group 2: PF--06473871/Placebo (3* 5 mg/cm)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated at the discretion of sponsor as study B5301001 did not meet its pre-defined efficacy endpoints for the dosing regimens evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.